CLINICAL TRIAL: NCT07111572
Title: Dynamic Changes of Fecal Calprotectin and Fecal Immunochemical Test for Early Prediction of Biologic Treatment Efficacy in Ulcerative Colitis: A Multicenter, Prospective Cohort Study
Brief Title: Fecal biOmarker Response Evaluation for Super-Early Efficacy in Ulcerative Colitis
Acronym: FORESEE-UC
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Qilu Hospital of Shandong University (Qingdao) (Other); Dezhou Hospital Qilu Hospital of Shandong University (Other); Weihai Municipal Hospital (Other); Liaocheng People's Hospital (Other); Jining First People's Hospital (Other)
Responsible Party: Principal Investigator, zhangyan, M.D, Qilu Hospital of Shandong University
Other Study IDs: QILUGI-003
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis (UC); Fecal Calprotetin; FIT
Keywords: UC; fecal calprotectin; FIT
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UC patients accept therapy of biologics
  Interventions: Diagnostic Test: fecal calprotectin

INTERVENTIONS:
Diagnostic Test: fecal calprotectin — patients will accpet test of FC combine FIT

SUMMARY:
This multicenter prospective cohort aims to evaluate whether combined changes in fecal calprotectin (FC) and fecal immunochemical test (FIT) at **Week 2 and Week 4** after initiating biologic therapy (vedolizumab or infliximab) can predict clinical response at **Week 14** and mucosal healing at **Week 52** in moderate-to-severe ulcerative colitis (UC) patients. Primary outcome: clinical remission rate at Week 14.

ELIGIBILITY:
Inclusion Criteria:**

* Age 18-75 years, UC diagnosis with endoscopic Mayo score (MES) ≥2
* Moderate-to-severe activity (Full Mayo Score ≥6)
* Initiating vedolizumab or infliximab within 7 days after baseline
* Biologic-naïve or prior exposure to only one TNF-α inhibitor

**Exclusion Criteria:**

* Pregnancy/lactation
* Contraindications to biologics (e.g., active TB, severe infection)
* Experimental drug use within 4 weeks prior to baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UC patinets accept biologics
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion achieving **clinical remission** (Full Mayo Score ≤2, no subscore >1) at **Week 14** | WEEK 14

SECONDARY OUTCOMES:
Mucosal healing (MES=0) at W52 | week 52
  Clinical response rate (W14)
  * Endoscopic improvement (MES ≤1) at W14
  * Steroid-free clinical remission at W52
  * Mucosal healing (MES=0) at W52
  * ROC analysis of FC/FIT for predicting outcome

IPD SHARING:
Plan to Share IPD: Undecided